CLINICAL TRIAL: NCT06592508
Title: Evaluation Of A Virtual Cardiology Program To Improve Outcomes After Acute Decompensated Heart Failure: The ELEVATE-HF Randomized Controlled Trial
Brief Title: Evaluation Of A Virtual Cardiology Program To Improve Outcomes After Acute Decompensated Heart Failure
Acronym: ELEVATE-HF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Ventricle Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00115672
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; With Decompensation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Remote Virtual Cardiology Program (Experimental): The Ventricle Health program will remotely receive daily vital signs directly from a blood pressure cuff and scale provided to the participant. In addition, the program will also remotely receive oxygen levels and electrical heart activity directly from a Pulse Ox and an EKG Single-Lead monitor, provided to the participant. All of this data will be transmitted to the Ventricle Health program. The Ventricle Health team, consisting of Cardiologists and clinical staff, will use this data to titrate medications and make clinical decisions.
  Interventions: Other: Remote Virtual Cardiology Program
- Usual Care (No Intervention): Routine clinical care will be followed. Participants should be recommended for the best possible outpatient heart failure care at each site.

INTERVENTIONS:
Other: Remote Virtual Cardiology Program — Ventricle Health Program, which is a remote, virtual, cardiology program that provides heart failure education to patients, monitors for worsening heart failure, and rapidly titrates heart failure medical therapy.
  Arms: Experimental: Remote Virtual Cardiology Program

SUMMARY:
The purpose of this study is to evaluate how safe and effective a remote, virtual, cardiology program is that provides heart failure education to patients, monitors for worsening heart failure, and quickly adjusts heart failure medications, compared to usual care medication use and adjustment, in participants with decompensated heart failure that are recently hospitalized.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age
* Acute decompensated HF as a primary cause of hospitalization. Hospitalizations for acute decompensated HF will be determined by local clinician-investigators but should include findings of acute HF (i.e., symptoms, signs, and/or laboratory/imaging abnormalities) and treatments aimed at acute HF (e.g., intravenous diuretics, vasodilators, or inotropes). Participants with a new diagnosis of HF may be enrolled. The enrollment will be monitored to ensure no more than 2/3 of the total cohort has new-onset HF.
* Fluent in written and spoken English

Exclusion Criteria:

* Optimized or nearly optimized on evidence-based medical therapies for HF as determined by local investigator
* Current pregnancy
* Chronic use of intravenous inotropic medications including milrinone, dobutamine, or dopamine
* eGFR of <20 mL/min/1.73m2 ongoing chronic dialysis at screening. The eGFR should be estimated using the 2021 Chronic Kidney Disease Epidemiology Collaboration (2021 CKD-EPI) creatinine equation.
* History of prior heart transplant or currently listed for heart transplant
* Current left ventricular assist device or planned left ventricular assist device in the next 6 months
* Currently receiving hospice care
* Chronically resides in an assisted living or skilled nursing facility where medications are managed by facility personnel
* Terminal illness other than HF with a life expectancy of <1 year as determined by the enrolling clinician-investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Time to all-cause death | Up to 120 days
Number of participants with worsening Heart Failure events | Up to 120 days
Time to first worsening Heart Failure event | Up to 120 days
Change in the number of classes of Heart Failure medications | Up to 120 days

SECONDARY OUTCOMES:
Number of participants with any intensification (initiation or dose titration) of evidence-based medical therapies for HF (heart failure) | Baseline, 120 days
Cumulative number of intensifications of evidence-based medical therapies for HF (heart failure) | Baseline, 120 days
Change in the number of classes of HF (heart failure) medications | Baseline, 120 days
  by different HF classifications as defined by LVEF
Composite of all-cause death and total worsening HF (heart failure) events defined by hospitalizations for acute decompensated HF and other urgent medical care for worsening HF | 30 day, 60 day, 120 day
Number of participants with combined Emergency department visits and hospitalizations | 30 day, 60 day, 120 day
  Combined Emergency department visits and hospitalizations related to evidence-based medical therapies for HF including symptomatic hypotension, hyperkalemia, and angioedema.

OTHER OUTCOMES:
Change in participant-reported medication adherence using the Voils score | Baseline, 120 day
  The Voils score includes questions used to assess medication adherence. Answers range between "not at all" and "very much", with 3 options in between. "Not at all" means a dose was not missed and "Very much" means dose was missed for that reason.
Change in Kansas City Cardiomyopathy Questionnaire Overall Summary score | Baseline, 120 day
  The Kansas City Cardiomyopathy Questionnaire 12-item version includes multiple domains: symptom frequency, quality of life, social limitation, and physical limitation. The Overall Summary score incorporates the averages of these 4 domains and is reported on a 0-to-100-point scale, where lower scores represent more severe symptoms and/or limitations and scores of 100 indicate no symptoms, no limitations, and excellent quality of life.
Net promoter score as assessed by the Ventricle Health Performance Survey | 120 day
Number of participants with All-cause hospitalization | 30 day, 60 day, 120 day

CONTACTS AND LOCATIONS:
Overall Officials: Adam DeVore, Principal Investigator — Duke University
Locations (5):
- United States (5):
  - Cardiovascular Institute of Northwest Florida, Panama City, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Premier Health, Dayton, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio

IPD SHARING:
Plan to Share IPD: No